CLINICAL TRIAL: NCT06978764
Title: Low Intensity Focused Ultrasound Modulation of Thalamic Nuclei for Central Neuropathic Pain: A Double- Blind Controlled Study.
Brief Title: Low Intensity Focused Ultrasound Modulation of Thalamic Nuclei for Central Neuropathic Pain.
Acronym: Thalamic LIFUP
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Ricardo de Carvalho Nogueira, Principal Investigator, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 35818919600000068
Record Dates: First submitted 2025-04-10; First posted 2025-05-18 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Central Neuropathic Pain
Keywords: plexo braquial

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active (Active Comparator): Patients receiveing Thalamic LIFUP intervention
  Interventions: Procedure: Thalamic LIFUP
- Sham (Sham Comparator): Patients receiveing Thalamic Sham intervention
  Interventions: Procedure: Thalamic LIFUP

INTERVENTIONS:
Procedure: Thalamic LIFUP — Patients will receive intervention in Thalamus region by LIFUP

SUMMARY:
LIFUP may have a modulatory effect on neuronal circuitry involved in pain, specifically when applied to the anterior thalamic nuclei, which is an important part of the pain circuit .Precise laboratory studies will reveal the indications under which LIFUP produces analgesia. The first step in evaluating LIFUP as a therapy for pain control is to determine whether LIFUP produces analgesia through suppression of the anterior thalamus. The primary objective is to evaluate the short-term analgesic effects of thalamic analgesia caused by LIFUP through:

1. Quantitative sensory testing (QST) and conditioned pain modulation testing (CPM) that allow the assessment of perceptual responses to quantifiable sensory stimuli, evaluated to characterize somatosensory function or dysfunction.
2. Short-form McGill Pain Questionnaire;
3. Brief Inventory Form, which includes pain severity index (average of questions 3-6) and pain interference with daily activities (average of questions 9A-9G, ranging from 0 to 70, where 70 indicates maximum possible pain interference);
4. Douleur Neuropathique-4 to assess neuropathic pain, being positive for scores ≥4;
5. Neuropathic Pain Symptom Inventory (NPSI), which provides characterization of neuropathic pain symptoms in 5 domains (superficial and deep) spontaneous pain, paroxysmal pain, evoked pain and paresthesia.

In association, analysis of its responses with others qualitative scales will be made described above:

1. Hamilton D + A
2. Medication use (Brief Pain Inventory)
3. Interference with daily activities (Brief Pain Inventory, quantified by Medication Quantification Scale)
4. Cognition - Montreal Cognitive Assessment (Mo CA)5 Adverse events
5. Blinding assessment
6. Variation in Global Impression of Change (CGI)

DETAILED DESCRIPTION:
Chronic pain (CP) is highly prevalent worldwide and has been identified as a major public health problem in many countries (1), being one of the ten leading causes of years lived with disability. CP has recently been identified as even more prevalent in countries with low human development indices (2-3). Pain affects 20-40% of the general population in Latin America and constitutes a major public health challenge (4-7). CP has known associations with depressed mood, fatigue, and catastrophic thinking. It is also widely recognized that even for CP directly triggered by peripheral structures, such as joints and muscles, there is a wide range of central changes (spinal cord, brain) occurring in CP, leading to a series of central modifications that will allow perpetuation and maintenance of the CP status (8-10). Pain is linked to maladaptive plasticity in the central nervous system (CNS) (8, 11-16), and structural and functional changes observed in the CNS during CP are related to symptom severity.

Central neuropathic pain (CNP) is caused by injury or disease of the somatosensory pathways in the CNS. CNP is a secondary complication of common diseases such as stroke (i.e., central post-stroke pain [CPSP]) and spinal cord injury (SCI) secondary to traumatic, inflammatory, or demyelinating diseases. CPSP occurs in 2% to 8% of stroke survivors and is present in up to 18% of those with somatosensory deficits and in up to 50% of those with lesions affecting only the spinothalamic pathways (20). Pain is also among the most debilitating complications of traumatic SCI (21), affecting more than 80% of patients within 5 years of trauma and leading to CNP in up to 59% of individuals. SCI It can also be caused by inflammatory insults that occur in demyelinating disorders such as multiple sclerosis (MS) or neuromyelitis optica spectrum disorders. These conditions affect more than 2 million individuals worldwide, leading to a lifetime prevalence of CNP of at least 28%. Unfortunately, attempts to control CNP have been marked by refractoriness and failure. For example, CPSP failed to respond satisfactorily to levetiracetam (22), pregabalin (23), duloxetine (24), morphine, and carbamazepine (25); while IBS-CNP did not respond to venlafaxine (26), levetiracetam (27), or dronabinol (28). MS-related CNP did not respond to cannabinoids (11) and duloxetine (29). In the rare positive trials that have existed, the magnitude of the analgesic effect has often been small, such as the response of CPSP/SCI-related CNP to duloxetine or pregabalin (30), or the response to opioids (31) in SCI-CNP. In other cases, positive results have been derived from very small studies. Thus, the treatment of CNP remains a major unmet need and has been the focus of several new treatment options, such as noninvasive neuromodulation.

The hallmark of CNP is the presence of pain with neuropathic descriptors in an area of impaired somatosensory function, often affecting thermal sensations (32). It has been proposed that damage to the spinothalamic projections would lead to plastic changes in brain areas implicated in pain processing; differentiation of insular pain receptors, leading to isolated functional disinhibition; and increased activity, causing increased processing of ascending stimuli by mesial pain pathways, including those targeting the parabrachial nucleus, anterior cingulate cortex (ACC) (33), and amygdala.

Although some aspects of this model have been questioned, the idea of an over-activation of these deep structures has been supported by functional brain imaging studies in normal humans in acute pain as well as in patients with neuropathic pain (34). Similarly, functional connectivity studies (35) have also reported a central role of these structures in neuropathic pain.

Low-intensity pulsed focused ultrasound (LIFUP) is a novel medical technology platform capable of neuromodulating regions of interest in the brain with high precision. Recent studies have shown LIFUP to be a safe and effective means of neuromodulation in pathologies such as trauma and epilepsy (36-37). Furthermore, focused ultrasound has been shown to induce reversible physiological effects on the nervous system, ranging from increased excitation in regions of interest to suppression of visual evoked potentials (38-39). Importantly, previous studies have observed both excitation and inhibition of neuronal circuits without characteristic physiological changes within the area of focus, such as cavitation or heat damage (40-44). Extrapolating from previous studies, LIFUP may have a modulatory effect on neuronal circuitry involved in pain, specifically when applied to the anterior thalamic nuclei, which is an important part of the pain circuitry (45). Precise laboratory studies will reveal the circumstances under which LIFUP produces analgesia. The first step in evaluating LIFUP as a therapy for pain management is to determine whether LIFUP produces analgesia through suppression of the anterior thalamus. Neurosurgical lesioning of the anterior thalamus has been used for many years as an invasive and risky treatment for this pain.

The primary objective is to evaluate the short-term analgesic effects of thalamic analgesia caused by LIFUP through:

1. Quantitative sensory testing (QST) and conditioned pain modulation testing (CPM) that allow the assessment of perceptual responses to quantifiable sensory stimuli, evaluated to characterize somatosensory function or dysfunction.
2. Short-form McGill Pain Questionnaire;
3. Brief Inventory Form, which includes pain severity index (average of questions 3-6) and pain interference with daily activities (average of questions 9A-9G, ranging from 0 to 70, where 70 indicates maximum possible pain interference);
4. Douleur Neuropathique-4 to assess neuropathic pain, being positive for scores ≥4;
5. Neuropathic Pain Symptom Inventory (NPSI), which provides characterization of neuropathic pain symptoms in 5 domains (superficial and deep) spontaneous pain, paroxysmal pain, evoked pain and paresthesia.

In association, analysis of its responses with others qualitative scales will be made described above:

1. Hamilton D + A
2. Medication use (Brief Pain Inventory)
3. Interference with daily activities (Brief Pain Inventory, quantified by Medication Quantification Scale)
4. Cognition - Montreal Cognitive Assessment (Mo CA)5 Adverse events
5. Blinding assessment
6. Variation in Global Impression of Change (CGI).

ELIGIBILITY:
Inclusion Criteria:

* Male or female more than 18 years old;
* Persistent presence of pain from braquial plexopathy injury for more than 3 months with an average of pain scoring of four or more points in numeric verbal scale (refractory to treatments).

Exclusion Criteria:

* history of uncontrolled epilepsy
* history of depression
* surgery or hospitalizations in the last 6 months
* presence of metal brain implants
* history of alcohol or drug addiction
* pregnancy
* history of loss of consciousness lasting more than 15 minutes

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-11-19 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-04-25 (Estimated)

PRIMARY OUTCOMES:
Pain assessments | Before and immediately after intervention. Also 4 hours, 24 hours, 10 days and 28 days after intervention.
  Pain scores in Visual Analog Scale has a numeric scoring that measures the intensity of pain from a scale of 1 to 10. The higher numeric scoring of the scale suggests severity and worse pain sensations.
  The scale will be analyzed before and after application of low-intensity pulsed ultrasound on the anterior thalamus.

SECONDARY OUTCOMES:
Somatosensory system analysis | Before intervention as well as immediately after and 28 days after intervention
  Change in somatosensory system will be evaluated by Quantitative Sensory Testing to identify perception of different sensory stimulus ( thermal and mechanical) before and after intervention. This is an individualized comparison assessment of each participant.

OTHER OUTCOMES:
Conditioned Pain Modulation | Before and immediately after intervention and after 28 days after intervention.
  Tests of Conditioned Pain Modulation will be analyzed to analyze endogenous pain inhibitory system. This is an individualized comparison assessment of each participant.
Neuropathic pain assessment | Before intervention as well as immediately after and 28 days after intervention
  Neuropathic Pain Symptom Inventory questionnaire will be assessed to understand severity, location and quality of participants pain. This is a scale that analyses from 1 to 10 . When the scale score achieve number 10, participants describes severity and worse pain sensations.
Depression and Anxiety analysis | Before and after 28 days of intervention.
  Change from baseline in Hamilton Depression Rating Scale and Anxiety ( HAM D/E) score after 28 days after intervention. The scale consist of 17 items ( rated by 0 to 4) and above 25 suggests severe depression.
Pain assessment in daily life | Before, immediately after and 28 days after intervention.
  As for understand pain impacts in daily life and severity, The Brief Pain Inventory (BPI) questionnaire will be assessed. It has a numeric rating scale for pain interference in activities. This is a 0 to 10 scale while score of 10 suggests severity of pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Neurology Department HCFMUSP, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ab Aziz CB, Ahmad AH. The role of the thalamus in modulating pain. Malays J Med Sci. 2006 Jul;13(2):11-8. PMID 22589599
- [Background] Monna T, Kuroki T, Oka H, Yamamoto S, Murata R, Suyama I, Issiki G, Nakao M. Prevention of vertical transmission of HBV by administration of hepatitis B vaccine combined with HBIG and long-term follow-up of HBsAb titer. Osaka City Med J. 1988 Jul;34(1):9-17. No abstract available. PMID 3419810
- [Background] Cruccu G, Garcia-Larrea L, Hansson P, Keindl M, Lefaucheur JP, Paulus W, Taylor R, Tronnier V, Truini A, Attal N. EAN guidelines on central neurostimulation therapy in chronic pain conditions. Eur J Neurol. 2016 Oct;23(10):1489-99. doi: 10.1111/ene.13103. Epub 2016 Aug 11. PMID 27511815
- [Background] Attal N, Ayache SS, Ciampi De Andrade D, Mhalla A, Baudic S, Jazat F, Ahdab R, Neves DO, Sorel M, Lefaucheur JP, Bouhassira D. Repetitive transcranial magnetic stimulation and transcranial direct-current stimulation in neuropathic pain due to radiculopathy: a randomized sham-controlled comparative study. Pain. 2016 Jun;157(6):1224-1231. doi: 10.1097/j.pain.0000000000000510. PMID 26845524
- [Background] Finnerup NB, Haroutounian S, Kamerman P, Baron R, Bennett DLH, Bouhassira D, Cruccu G, Freeman R, Hansson P, Nurmikko T, Raja SN, Rice ASC, Serra J, Smith BH, Treede RD, Jensen TS. Neuropathic pain: an updated grading system for research and clinical practice. Pain. 2016 Aug;157(8):1599-1606. doi: 10.1097/j.pain.0000000000000492. PMID 27115670
- [Background] Peyron R, Laurent B, Garcia-Larrea L. Functional imaging of brain responses to pain. A review and meta-analysis (2000). Neurophysiol Clin. 2000 Oct;30(5):263-88. doi: 10.1016/s0987-7053(00)00227-6. PMID 11126640
- [Background] de Oliveira RA, de Andrade DC, Machado AG, Teixeira MJ. Central poststroke pain: somatosensory abnormalities and the presence of associated myofascial pain syndrome. BMC Neurol. 2012 Sep 11;12:89. doi: 10.1186/1471-2377-12-89. PMID 22966989
- [Background] Hosomi K, Shimokawa T, Ikoma K, Nakamura Y, Sugiyama K, Ugawa Y, Uozumi T, Yamamoto T, Saitoh Y. Daily repetitive transcranial magnetic stimulation of primary motor cortex for neuropathic pain: a randomized, multicenter, double-blind, crossover, sham-controlled trial. Pain. 2013 Jul;154(7):1065-72. doi: 10.1016/j.pain.2013.03.016. Epub 2013 Mar 15. PMID 23623156
- [Background] Kim JS, Bashford G, Murphy KT, Martin A, Dror V, Cheung R. Safety and efficacy of pregabalin in patients with central post-stroke pain. Pain. 2011 May;152(5):1018-1023. doi: 10.1016/j.pain.2010.12.023. Epub 2011 Feb 12. PMID 21316855
- [Background] Jungehulsing GJ, Israel H, Safar N, Taskin B, Nolte CH, Brunecker P, Wernecke KD, Villringer A. Levetiracetam in patients with central neuropathic post-stroke pain--a randomized, double-blind, placebo-controlled trial. Eur J Neurol. 2013 Feb;20(2):331-7. doi: 10.1111/j.1468-1331.2012.03857.x. Epub 2012 Aug 27. PMID 22925226
- [Background] Siddall PJ, McClelland JM, Rutkowski SB, Cousins MJ. A longitudinal study of the prevalence and characteristics of pain in the first 5 years following spinal cord injury. Pain. 2003 Jun;103(3):249-257. doi: 10.1016/S0304-3959(02)00452-9. PMID 12791431
- [Background] Vartiainen N, Perchet C, Magnin M, Creac'h C, Convers P, Nighoghossian N, Mauguiere F, Peyron R, Garcia-Larrea L. Thalamic pain: anatomical and physiological indices of prediction. Brain. 2016 Mar;139(Pt 3):708-22. doi: 10.1093/brain/awv389. Epub 2016 Feb 8. PMID 26912644